CLINICAL TRIAL: NCT02217228
Title: A Randomized, Prospective, Multicenter, Controlled Study With Blinded Assessment to Determine the Safety and Effectiveness of the Sebacia Acne Treatment System in the Treatment of Inflammatory Acne Vulgaris
Brief Title: Pivotal Study of Sebacia Microparticles in the Treatment of Acne Vulgaris
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sebacia, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SEB-0121; IDE #G120273 (Other: FDA CDRH)
Record Dates: First submitted 2014-08-11; First posted 2014-08-15 (Estimated); Last update posted 2017-09-18 (Actual); Status verified 2017-09

CONDITIONS: Inflammatory Acne Vulgaris
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sebacia microparticles and laser (Experimental): Gold microparticle suspension + laser treatment x 3 over the course of two weeks
  Interventions: Device: Sebacia microparticles and laser
- Vehicle suspension and laser (Experimental): Vehicle suspension + laser treatment x 3 over the course of two weeks
  Interventions: Device: Vehicle suspension and laser
- Sebacia microparticles without laser (Experimental): Gold microparticle suspension treatment x 3 over the course of two weeks
  Interventions: Device: Sebacia microparticles without laser

INTERVENTIONS:
Device: Sebacia microparticles and laser
  Arms: Sebacia microparticles and laser
Device: Vehicle suspension and laser
  Arms: Vehicle suspension and laser
Device: Sebacia microparticles without laser
  Arms: Sebacia microparticles without laser

SUMMARY:
Prospective, randomized multicenter study to examine the safety and effectiveness of Sebacia microparticles with or without laser in the treatment of moderate to moderately-severe inflammatory acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 15 - 45 years of age
* Able to provide informed consent/assent; minors will provide assent while parent or legal guardian will provide consent
* Moderate to moderately severe (3 or 4) inflammatory acne vulgaris by Investigator's Global Assessment
* Subject has 25 to 75 inflammatory lesions on the cheeks, chin and forehead, not concentrated in one area
* Subject has Fitzpatrick skin phototype I, II or III
* Subject is in good health, willing to participate and able to comply with protocol requirements

Exclusion Criteria:

* Severe acne (Investigator's Global Assessment 5) with significant scarring potential and greater than 2 nodular lesions
* Clinically relevant history of keloids
* Facial tattoos
* Acne conglobata, acne fulminans, chloracne, drug-induced acne
* Active concomitant skin disease, excessive scarring or excess facial hair
* Heavily tanned skin; unable or unwilling to avoid tanning beds/excessive sun exposure
* Acne medication and therapy restrictions - time period prior to Baseline (below)

  1. Oral retinoids - 6 months
  2. Other systemic medications - 4 weeks
  3. Topical retinoids, steroids, antibiotics - 2 weeks
  4. OTC topical treatments - 1 week
  5. Light treatments (including IPL or laser), microdermabrasion and/or peels - 8 weeks
  6. Investigational drug, biologic or device - 30 days
  7. Gold therapy of any type for any reason - EXCLUDED
* Pregnant, lactating, nursing or planning to become pregnant during the study period
* Known allergy to gold, ethanol, diisopropyl adipate, Polysorbate 80
* Clinically relevant condition that makes participation unsafe or that would interfere with study treatment and assessment

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 394 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Mean percent change in inflammatory lesion count from Baseline to Week 12 | Week 12
Number of of adverse events | Screening to 12 Weeks

SECONDARY OUTCOMES:
Mean absolute change in inflammatory lesion count from Baseline to Week 12 | Week 12
Success by Investigator's Global Assessment at Week 12 (defined as 2-point decrease from Baseline IGA) | Week 12

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Clear Dermatology & Aesthetics Center, Scottsdale, Arizona
  - Laser & Skin Surgery Center of Northern California, Sacramento, California
  - Center for Dermatology & Laser Surgery, Sacramento, California
  - Miami Dermatology & Laser Institute, Miami, Florida
  - Spencer Dermatology, St. Petersburg, Florida
  - Gwinnett Dermatology, PC, Snellville, Georgia
  - The Dermatology Institute-DuPage Medical Group, Naperville, Illinois
  - Shideler Clinical Research Center, Carmel, Indiana
  - Maryland Laser, Skin & Vein Institute, Hunt Valley, Maryland
  - Clarkston Skin Research, Clarkston, Michigan
  - James Q Del Rosso, DO, LLC, Las Vegas, Nevada
  - Skin Laser & Surgery Specialists of NY & NJ, Hackensack, New Jersey
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Yardley Dermatology Associates, Yardley, Pennsylvania
  - Dermatology & Laser Center of Charleston, Charleston, South Carolina
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Austin Institute for Clinical Research, Pflugerville, Texas
  - Spokane Dermatology Clinic, Spokane, Washington